CLINICAL TRIAL: NCT02944760
Title: Acute Effects of Low-level Laser Therapy in Functional Capacity of Patients With Chronic Kidney Disease: Randomized Clinical Trial
Brief Title: Low-level Laser Therapy in Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLLT/CKD
Record Dates: First submitted 2016-10-11; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-Level Light Therapy Group (Experimental): The patient was placed supine on a stretcher and the application will take place with the Chattanooga device, with the laser diode cluster probe from the same manufacturer consisting of five diodes 850 nm and power output of 200 mW. Six points in quadriceps and four points in gastrocnemius, were irradiated, bilaterally, by 30 seconds.
  Interventions: Other: Low-Level Light Therapy
- Placebo Group (Placebo Comparator): The patient was placed supine on a stretcher and the application of laser therapy occured with apparatus off.
  Interventions: Other: Low-Level Light Therapy

INTERVENTIONS:
Other: Low-Level Light Therapy — The application of laser therapy will take place 30 minutes before the start of dialysis. The application will take place with the Chattanooga device, with the laser diode cluster probe from the same manufacturer consisting of five diodes 850 nm and power output of 200 mW. It is irradiated 6 points in quadriceps and 4 points in gastrocnemius, bilaterally by 30 seconds. The patient will be supine on a stretcher to the implementation of the intervention.
  Other Names: Laser Therapy, Low-Level

SUMMARY:
Chronic kidney disease is a renal injury and progressive and irreversible loss of kidney function and in its most advanced stage is called chronic renal failure. Although hemodialysis replace some kidney function, patients suffer some alterations characterized by "uremic syndrome" typically expressed by: motor neuropathy and/or autonomic neuropathy, cardiac or musculoskeletal myopathies, peripheral vascular changes, among others. Thus, the functional capacity and ability to exercise presents diminished these patients. The aim of this study is to verify the acute effect of low level laser therapy on the functional capacity of these individuals.

The research will be developed in the hemodialysis unit of the Santa Clara hospital of Santa Casa de Misericordia de Porto Alegre and the patients will be evaluated before and immediately after the application of laser therapy protocol. Before the protocol will be evaluated pain in the lower limbs, Borg scale, level of physical activity through the International Physical Activity Questionnaire (IPAQ) and blood collection will be held for later analysis parameters of biochemical oxidative stress and deoxyribonucleic acid (DNA) damage.

The laser therapy protocol will be applied in 6 points in quadriceps and 4 points in the gastrocnemius, bilaterally. After application, will be held the 6-minute walk test, effort subjective perception by Borg scale, assessment of pain in the lower limbs with visual analog scale and a new blood sample for further analysis. Patients will be randomized in two groups. The intervention group (IG), which will be held laser therapy and placebo group (PG), where the laser therapy will be placebo mode applied. The application will take place with the Chattanooga device, with the laser diode cluster probe from the same manufacturer consisting of five diodes 850 nanometers (nm) and power output of 200 milliwatts (mW). It is irradiated 6 points in quadriceps and 4 points in gastrocnemius, bilaterally.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease on hemodialysis for more than 3 months;
* Clearance of urea during hemodialysis (Kt/V ≥ 1.2).

Exclusion Criteria:

* Cognitive impairment that prevents conducting evaluations, as well as inability to understand and sign the informed consent form;
* Epidermal lesions at the site of application and/or intolerance stimulator and/or skin sensitivity change;
* Patients with recent sequel of stroke;
* Disabling musculoskeletal disease;
* Uncontrolled hypertension (Systolic blood pressure > 230 mmHg and diastolic blood pressure > 120 mmHg);
* Grade IV heart failure (NYHA) or decompensated;
* Uncontrolled diabetes (blood glucose > 300 mg/dL);
* Unstable angina;
* Fever and/or infectious disease;
* Recent acute myocardial infarction (two months);
* Active smokers; Peripheral vascular disease in the lower limbs as deep vein thrombosis or obliterates thromboangiitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | 15 minutes after intervention
  Assessed by the change in distance walked in six-minute walk test (6MWT)

SECONDARY OUTCOMES:
Pain in lower limbs | 15 minutes after intervention and 15 minutes after of 6MWT
  Assessed by change in visual analog scale
Dyspnea | 15 minutes after intervention and 15 minutes after of 6MWT
  Assessed by change in Borg scale
Level of physical activity | 30 minutes before of intervention
  Assessed by questionnaire IPAQ.
Oxidative stress will be assessed through blood collection and analysis of biochemical markers, such as creatine kinase, lactate and Oxygen-reactive species | 30 minutes before and 30 minutes after intervention
  Analysis of changes in biochemical markers, such as creatine kinase, lactate and oxygen-reactive species
DNA damage | 30 minutes before and 30 minutes after intervention
  By electrophoresis single (comet technique), where cells are counted by microscopy and and the breaks will be checked

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre

IPD SHARING:
Plan to Share IPD: Yes